CLINICAL TRIAL: NCT05396586
Title: Assessment and Training of Cognitive Function
Brief Title: Understanding Individual Differences in Working Memory Training and Transfer in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Collaborators: University of California, Riverside (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Susanne Jaeggi, Assistant Project Scientist, Northeastern University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 20141547; 1R21AG069428-01A1 (NIH); 5R21AG069428-02 (NIH)
Record Dates: First submitted 2022-04-21; First posted 2022-05-31 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-01

CONDITIONS: Cognitive Change

STUDY DESIGN:
Intervention Model Description: Three randomized crossover trials (N-back, Span and Multisensory) will be conducted and in each trial, participants will be randomly assigned to 1 of 2 conditions: Condition 1 consists of training type 1 followed by training type 2, whereas Condition 2 consists of training type 2 followed by training type 1. In the N-back trial, participants will be assigned to Non-Gamified N-back training and Gamified N-back training. In the Span trial, they will be assigned to Non-Gamified Span training and Gamified Span training and in the Multisensory trial, they will be assigned to Non-gamified Unisensory N-back training and Non-gamified Multisensory N-back training.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Condition 1 (Active Comparator): Training type 1 will be administered in the first part of the crossover trial and Training type 2 will be administered in the second part of the trial. Each training part consists of 20 twenty-minute long sessions with the recommended frequency of 2 sessions per work day. Thus each training part can be completed in 10 work days (2 weeks).
  Interventions: Behavioral: N-back; Behavioral: Span; Behavioral: Multisensory
- Condition 2 (Active Comparator): Training type 2 will be administered in the first part of the crossover trial and Training type 1 will be administered in the second part of the trial. Each training part consists of 20 twenty-minute long sessions with the recommended frequency of 2 sessions per work day. Thus each training part can be completed in 10 work days (2 weeks).
  Interventions: Behavioral: N-back; Behavioral: Span; Behavioral: Multisensory

INTERVENTIONS:
Behavioral: N-back — The training program is a personal device-based adaptive version of a visual N-back task, either devoid of game elements or embedded in a gamified platform game
Behavioral: Span — The training program is a personal device-based adaptive version of a visual working memory span task, either devoid of game elements or embedded in a gamified platform game
Behavioral: Multisensory — The training program is a personal device-based adaptive version of an N-back task that features visual stimuli (Unisensory) or visual stimuli paired with unique sounds (Multisensory) and is devoid of game elements

SUMMARY:
The present study investigates how individual differences in cognitive processing contribute to the efficacy of working memory training programs in an older adult population. In a randomized crossover design, different types of working memory training interventions will be evaluated within the same participants.

Adding game-like elements to working memory training programs can increase motivation and engagement, which can increase learning. However this process, termed gamification, adds sensory complexity that can lead to increased mental load and/or distraction in older adults. Investigators hypothesize that gamification of training tasks will be beneficial to some and counterproductive to other participants. The investigators will test two models; the first assumes that participants with difficulty inhibiting distracting information will show better learning and transfer when assigned to non-gamified training, whereas those with more distractor tolerance will show better learning and transfer when assigned to gamified training. The second model states that the outcomes of the intervention will be better predicted by performance on measures of general cognitive ability.

In a separate study, the investigators will compare working memory training that contains rich, multisensory information with a training program that contains only visual information. Here they will also test two models; the first assumes that participants with difficulty binding two stimulus streams will show better learning and transfer when assigned to visual-only working memory training, whereas participants who do not have this difficulty will show better learning and transfer when assigned to multisensory working memory training. The second model states that the outcomes of the intervention will be better predicted by performance on measures of general cognitive ability.

DETAILED DESCRIPTION:
Three randomized cross-over trials will be conducted to obtain within-subject comparisons of training with enriched (game-like) versions of working memory training tasks compared to basic (non-gamified) versions of these tasks. In the N-back trial, participants will be assigned to Non-Gamified N-back training and Gamified N-back training. In the Span trial, they will be assigned to Non-Gamified Span training and Gamified Span training and in the Multisensory trial, they will be assigned to Non-gamified Unisensory N-back training and Non-gamified Multisensory N-back training.

Each trial involves a total of 50 sessions per participant: the first few sessions consist of completing questionnaires and computerized cognitive assessments (pre-test). Participants then complete 20 sessions of working memory training. After a mid-test, they complete 20 sessions of a different type of working memory training. Post-test is administered upon training completion, and at least a month later, participants complete 3 follow-up sessions. The study can be administered either in person or remotely; however, the investigators anticipate that most participants will complete the study remotely.

ELIGIBILITY:
Inclusion Criteria:

* 50-85 years of age
* Able to understand and speak English and follow study procedures
* Does not have a psychological or neurological condition that would prevent being able to give consent to participate
* Not currently involved in any other cognitive or memory training studies

Exclusion Criteria:

* Formal diagnosis of dementia or other neurological disease, including Mild cognitive impairment.
* A final total score below 17 on Montreal Cognitive Assessment - Blind (telephone) version.
* Score of 10 or more on the Generalized Anxiety Questionnaire (GAD7; Spitzer et al., 2006, Archives of Internal Medicine), indicating presence of moderate or severe anxiety
* Score of 9 or more on Geriatric depression scale (GDS15; Yesavage et al., 1982) indicating presence of moderate or severe depression
* Abnormal visual acuity prohibitive of tablet-based training.
* Physical handicap (motor or perceptual) that would impede training procedures.
* Medical illness requiring treatment and/or significant absences during the study timeline.
* Current evidence or 2-yr history of seizures, focal brain lesion, or head injury with loss of consciousness.
* Current alcohol consumption exceeds 14 drinks per week.
* Self-reported illicit drug use.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Change in N-level | Day 24, Day 46, Day 78
  N-back is a tablet-based updating working memory task. Participants see a consecutive stream of pictures and are asked to tap the pictures that match those presented N items earlier. All participants will complete 1-back and 2-back, progression to 3-back and beyond is based on performance on the previous level (no more than 4 errors). The outcome measure is the change in the highest N-level reached on the task compared to baseline at Day 2.
Change in Corsi span | Day 25, Day 47, Day 79
  Corsi is a tabled-based measure of spatial working memory. Participants see characters emerge one at a time from twelve possible locations and are asked to repeat the sequence by tapping on the locations in the correct order. The task starts with set size two and increases in difficulty using an adaptive algorithm. Participants first play Simple Corsi (without a distractor task), followed by Complex Corsi (with a distractor task). The outcome measure is change in overall span, calculated as the sum of the two highest set sizes that can be recalled in Simple and Complex Corsi tasks, at the point of measurement compared to baseline at Day 3.
Change in Inhibitory Control Composite Score | Day 24, Day 46, Day 78
  The score is the mean of standardized dependent variables on tablet-based inhibitory control tasks. The outcome measure is the change in the composite score at the point of measurement compared to baseline at Day 2.
Change in Everyday Memory Questionnaire Revised | Day 24, Day 46, Day 77
  The Everyday Memory Questionnaire Revised (Royle & Lincoln, 2008) consists of 13 items that describe everyday events that might involve forgetting. Participants are asked how often on average they think each one has happened to them over the past month on a 5-point scale (0-4) and the total score is calculated as the sum of all responses. The minimum total score is 0 and the maximum is 52, with higher scores indicative of greater presence of memory difficulties. The outcome measure is the change in total score at the point of measurement compared to baseline at Day 1.

SECONDARY OUTCOMES:
Training Experience Enjoyment Subscale I | Day 24
  Scores range from 1 to 5, with higher scores indicative of greater enjoyment of the training task.
Training Experience Enjoyment Subscale II | Day 46
  Scores range from 1 to 5, with higher scores indicative of greater enjoyment of the training task.
Training Experience Difficulty Subscale I | Day 24
  Score range from 1 to 10, with scores 1-3 indicating that the training was too easy, scores 4-7 indicating that the training was of appropriate difficulty, and scores 8-10 indicating that it was too difficult.
Training Experience Difficulty Subscale II | Day 46
  Score range from 1 to 10, with scores 1-3 indicating that the training was too easy, scores 4-7 indicating that the training was of appropriate difficulty, and scores 8-10 indicating that it was too difficult.
Training Experience Subjective Progress Subscale I | Day 24
  Scores range from 1 to 5, with higher scores indicative of greater subjective progress on the training task.
Training Experience Subjective Progress Subscale II | Day 46
  Scores range from 1 to 5, with higher scores indicative of greater subjective progress on the training task.
Training Experience Interface Subscale I | Day 24
  Scores range from 1 to 5, with higher scores indicative of greater satisfaction with the interface (software).
Training Experience Interface Subscale II | Day 46
  Scores range from 1 to 5, with higher scores indicative of greater satisfaction with the interface (software).
Exit Survey | Day 79
  Participants are asked 5 open-ended questions about their subjective experience of participating in the study.

OTHER OUTCOMES:
Change in General Cognitive Ability Composite Score | Day 77
  A composite score will be generated by taking the average of standardized outcome measures on tasks in the Standard Older Adult Cognitive Battery (SOACB), which consists of word list learning, complex figure copy, object naming, trail making, a vocabulary task, and matrix reasoning. The outcome measure is the change in the composite score reached on the task compared to baseline at Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron R Seitz, Phd, Principal Investigator — University of California, Riverside; Susanne M Jaeggi, Phd, Principal Investigator — University of California, Irvine
Locations (2):
- United States (2):
  - University of California, Irvine, Irvine, California
  - University of California, Riverside, Riverside, California

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (anonymized).
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available persistently at the conclusion of the study.
Access Criteria: There are no access criteria.

REFERENCES:
- [Background] Pahor A, Mester RE, Carrillo AA, Ghil E, Reimer JF, Jaeggi SM, Seitz AR. UCancellation: A new mobile measure of selective attention and concentration. Behav Res Methods. 2022 Oct;54(5):2602-2617. doi: 10.3758/s13428-021-01765-5. Epub 2022 Feb 1. PMID 35106729
- [Background] Pahor A, Stavropoulos T, Jaeggi SM, Seitz AR. Validation of a matrix reasoning task for mobile devices. Behav Res Methods. 2019 Oct;51(5):2256-2267. doi: 10.3758/s13428-018-1152-2. PMID 30367386
- [Background] Royle J, Lincoln NB. The Everyday Memory Questionnaire-revised: development of a 13-item scale. Disabil Rehabil. 2008;30(2):114-21. doi: 10.1080/09638280701223876. PMID 17852284
- [Background] Pahor A, Collins C, Smith RN, Moon A, Stavropoulos T, Silva I, Peng E, Jaeggi SM, Seitz AR. Multisensory Facilitation of Working Memory Training. J Cogn Enhanc. 2021 Sep;5(3):386-395. doi: 10.1007/s41465-020-00196-y. Epub 2020 Nov 27. PMID 34485810
- [Background] Sandeep S, Shelton CR, Pahor A, Jaeggi SM, Seitz AR. Application of Machine Learning Models for Tracking Participant Skills in Cognitive Training. Front Psychol. 2020 Jul 22;11:1532. doi: 10.3389/fpsyg.2020.01532. eCollection 2020. PMID 32793032